CLINICAL TRIAL: NCT03305198
Title: BIOlogical Response to Exercise : A Metabolomic Study in Peripheral Artery Disease (BIOR)
Acronym: BIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-A01147-46
Record Dates: First submitted 2017-09-28; First posted 2017-10-09 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Analysis of changes in metabolomic signature from rest to post exercise
Masking Description: Metabolomic analysis will be performed blinded to the exercise test results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing exercise oximetry (Experimental): Patients with PAD referred for treadmill testing and exercise oximetry will have a capillary blood sampling from the earlobe
  Interventions: Biological: Capillary blood sampling from the earlobe

INTERVENTIONS:
Biological: Capillary blood sampling from the earlobe — Sample at rest before the walking test Sample at rest 3 minutes after the end of the walking period

SUMMARY:
The measurement of the transcutaneous oxygen pressure during walking allows to estimate the importance of ischemia, bilaterally and segment of limb by segment of limb. The determination of the metabolic compounds concentration, with metabolomic approach, is emerging in physiology and exercise.

This pilot study focuses on the feasibility of the metabolomics analysis with micro method , by capillary drawing from earlobe sampling, for patients with peripheral artery disease (PAD)

DETAILED DESCRIPTION:
Ankle brachial index is measured at rest for alml subjects. Blood sample (180-360 microliter) will be collected at rest transcutaneous oxygen pressure is measured at the chest, calves and buttocks and results will be expressed as the minimal value of the DROP index (Limb changes minus chest changes) Patients walk on treadmill (2MPH 10% slope) until exertional limb pain. Blood sample (180 microliter) will be collected again, at minute 3 of recovery from walking Correlation of each metobolite increase to the sum of DROP values wil be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient able to walk on a treadmill
* Patient agrees to be involve in the protocol and sign the consent form

Exclusion Criteria:

* Patient not covered by the French health insurance
* Patient has a wash-out period for another clinical trial
* Patient with comorbidity as bleeding disorder or with a anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Chances in the metabolomic signature of arterial claudication by capillary blood sampling from the earlobe | Half an hour (includes the resting walking and recovery period of exercise)
  Search a significant difference between biological markers before and after the test during a walk on a treadmill

SECONDARY OUTCOMES:
Changes inthe correlation of observed metabolomic variations and the importance of ischemia evaluated by oximetry | Half an hour (includes the resting walking and recovery period of exercise)
  Evaluate the coefficient of correlation between the changes of metabolomic pârameters and the sum of the observed DROPmin values of all studied subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD, Ph.D, Principal Investigator — University Hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided